CLINICAL TRIAL: NCT02310256
Title: A Randomized Clinical Trial on the Effects of Home-based Five Plus Exercise Training
Brief Title: A Clinical Trial on the Effects of Home-based Five Plus Exercise Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011/2533/REK midt
Record Dates: First submitted 2014-11-10; First posted 2014-12-08 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Intermittent Claudication
Keywords: Mitochondria, muscle; Exercise; Blood Flow Velocity
MeSH Terms: conditions — Intermittent Claudication; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention)
- Five Plus (Active Comparator): Exercise training
  Interventions: Other: Five plus exercise training

INTERVENTIONS:
Other: Five plus exercise training — calf raise exercise
  Arms: Five Plus

SUMMARY:
The aim of the study is to evaluate whether walking capacity in patients with intermittent claudication is improved more by home-based 5+ exercise training than by current recommendations of daily walking. The study will elucidate if such a potential effect is dependent on changes in mitochondrial respiratory capacity, blood flow or both.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with intermittent claudication secondary to vascular insufficiency
* An ankle-brachial index between 0.4 and 0.9.

Exclusion Criteria:

* Diagnosed with critical limb ischemia
* Ankle-brachial index (ABI) > 0.90 or < 0.4
* Limited exercise tolerance
* Warfarin or heparin usage
* Underwent a vascular intervention in the last 6 months
* Active cancer, renal- or liver disease

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
absolute walking distance (meters) as measured by 6 minute walking test | 8 weeks
  treadmill 3.2 km/hour and inclination increase every 2 minute combined with 6 minute walking test
mitochondrial function measured by respirometry | 8 weeks
  Oxygen consumption (pmol O2 per second per mg of wet weight tissue) measured by respirometry

SECONDARY OUTCOMES:
Arterial bloodflow measured by plethysmography | 8 weeks
  measured by plethysmography
Quality of life assessed by SF 36 and CLAU-S questionnaires | 8 weeks
  assessed by SF 36 and CLAU-S questionnaires
Peak oxygen uptake measured by cardio-pulmonal exercise testing | 8 weeks
  measured by cardio-pulmonal exercise testing

CONTACTS AND LOCATIONS:
Overall Officials: Øivind Rognmo, phd, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department for circulation and medical imaging, NTNU, Trondheim, Postboks 8905, Norway

REFERENCES:
- [Result] Van Schaardenburgh M, Wohlwend M, Rognmo O, Mattsson E. Calf raise exercise increases walking performance in patients with intermittent claudication. J Vasc Surg. 2017 May;65(5):1473-1482. doi: 10.1016/j.jvs.2016.12.106. Epub 2017 Mar 9. PMID 28285932
- [Result] van Schaardenburgh M, Wohlwend M, Rognmo O, Mattsson EJR. Exercise in claudicants increase or decrease walking ability and the response relates to mitochondrial function. J Transl Med. 2017 Jun 7;15(1):130. doi: 10.1186/s12967-017-1232-6. PMID 28592294